CLINICAL TRIAL: NCT01016990
Title: Epigenetic Therapy With Valproic Acid, an HDAC Inhibitor, in Refractory/Relapsed Non-Hodgkin Lymphoma, Hodgkin's Disease and CLL
Brief Title: Valproic Acid in Treating Patients With Previously Treated Non-Hodgkin Lymphoma, Hodgkin Lymphoma, or Chronic Lymphocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000659192; CCAM-HDACI
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-11

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; recurrent cutaneous T-cell non-Hodgkin lymphoma; peripheral T-cell lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related lymphoblastic lymphoma; Waldenström macroglobulinemia
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Waldenstrom Macroglobulinemia | interventions — Valproic Acid; Blotting, Western

INTERVENTIONS:
Drug: valproic acid
Genetic: western blotting
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Valproic acid may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It may also help cancer cells become more like normal cells, and grow and spread more slowly.

PURPOSE: This phase II trial is studying how well valproic acid works in treating patients with previously treated non-Hodgkin Lymphoma, Hodgkin lymphoma, or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if valproic acid has a response rate of ≥ 20% in patients with previously treated relapsed or refractory non-Hodgkin lymphoma, Hodgkin lymphoma, or chronic lymphocytic leukemia.
* To determine if treatment with valproic acid leads to measurable levels of histone acetylation in peripheral blood.

OUTLINE: Patients are stratified according to disease diagnosis (indolent non-Hodgkin lymphoma [NHL] vs. aggressive NHL and Hodgkin lymphoma). Valproic acid doses are adjusted until therapeutic level is achieved.

Patients receive oral valproic acid daily for 3 weeks. Treatment repeats every 3 weeks for at least 2 courses and up to 2 years in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically. Samples are analyzed for valproic acid levels; and hyperacetylation (caused by the valproic acid N-terminals of the histones H3 and H4) via western blot.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory Hodgkin lymphoma (HL), non-Hodgkin lymphoma (NHL), or chronic lymphocytic leukemia (CLL )
* Patient must have evaluable or measurable disease
* Have failed prior treatment, as evidenced by 1 of the following:

  * Aggressive NHL

    * Failed at least 1 regimen containing rituximab and CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone) (unless anthracyclines are contraindicated) in addition to another salvage regimen (unless it is determined by the treating physician that it is to the patient's best interest to receive valproic acid after the first relapse)
  * Hodgkin lymphoma

    * Failed ABVD (doxorubicin, bleomycin, vinblastine, and dacarbazine) and received salvage chemotherapy with at least 1 salvage combination regimen
  * Indolent or low-grade lymphoma

    * Failed at least 1 combination regimen containing rituximab (patients who are intolerant to the available therapies or have contraindications for them are eligible for the study)
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,000/mm^3
* Platelet count ≥ 50,000/µL
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* More than 14 days since prior anticancer treatment
* Prior high-dose chemotherapy with transplant allowed
* No prior valproic acid
* No concurrent corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Response to therapy (complete response, partial response, or stable disease)

SECONDARY OUTCOMES:
Length of response
Time to treatment failure
Survival duration

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Auxilio Mutuo Cancer Center
Locations (1):
- Centro de Cancer del Hospital Auxilio Mutuo, San Juan, Puerto Rico